CLINICAL TRIAL: NCT06465576
Title: Strategy for Withdrawal of Pharmacological Treatment for Urinary Incontinence in Children (StayDry)
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: StayDry
Record Dates: First submitted 2024-06-13; First posted 2024-06-20 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Urinary Incontinence in Children
Keywords: Urinary incontinence; Withdrawal; Children; Solifenacin; Mirabegron
MeSH Terms: conditions — Urinary Incontinence | interventions — Solifenacin Succinate; mirabegron

STUDY DESIGN:
Intervention Model Description: Within each pharmaceutical group, the participant will be randomized 1:1 to the intervention being compared; either abrupt withdrawal or gradual withdrawal.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Abrupt withdrawal of solifenacin (Experimental)
  Interventions: Drug: Solifenacin
- Gradual withdrawal of solifenacin (Experimental)
  Interventions: Drug: Solifenacin
- Abrupt withdrawal of mirabegron (Experimental)
  Interventions: Drug: Mirabegron
- Gradual withdrawal of mirabegron (Experimental)
  Interventions: Drug: Mirabegron
- Abrupt withdrawal of solifenacin + mirabegron (Experimental)
  Interventions: Drug: Solifenacin + Mirabegron
- Gradual withdrawal of solifenacin + mirabegron (Experimental)
  Interventions: Drug: Solifenacin + Mirabegron

INTERVENTIONS:
Drug: Solifenacin — Abrupt withdrawal indicates stopping the medication on the date of withdrawal initiation.
  Gradual withdrawal involves taking the applied dosage of the medication every other day over a period of 14 days, with the complete cessation of the medication occurring 14 days after the gradual withdrawal process begins.
  Arms: Abrupt withdrawal of solifenacin; Gradual withdrawal of solifenacin
Drug: Mirabegron — Abrupt withdrawal indicates stopping the medication on the date of withdrawal initiation.
  Gradual withdrawal involves taking the applied dosage of the medication every other day over a period of 14 days, with the complete cessation of the medication occurring 14 days after the gradual withdrawal process begins.
  Arms: Abrupt withdrawal of mirabegron; Gradual withdrawal of mirabegron
Drug: Solifenacin + Mirabegron — Abrupt withdrawal indicates stopping the medication on the date of withdrawal initiation.
  Gradual withdrawal involves taking the applied dosage of the medication every other day over a period of 14 days, with the complete cessation of the medication occurring 14 days after the gradual withdrawal process begins.
  Arms: Abrupt withdrawal of solifenacin + mirabegron; Gradual withdrawal of solifenacin + mirabegron

SUMMARY:
The primary objective is to investigate if abrupt withdrawal versus gradual withdrawal of pharmacotherapy (solifenacin and/or mirabegron) influences the risk of recurrence of incontinence.

Children aged 5-14 years diagnosed with urinary incontinence, treated with pharmacotherapy of solifenacin and/or mirabegron and ready for withdrawal will be randomized 1:1 to either abrupt or gradual withdrawal, according to the medical treatment that the child is receiving.

DETAILED DESCRIPTION:
Background and rationale: The pharmacological handling of pediatric incontinence is considered temporary and withdrawal attempts are recommended after continence has been achieved. There is no generally accepted withdrawal strategy for solifenacin and/or mirabegron in children. Currently, two different withdrawal strategies are being employed in the clinical setting, namely abrupt withdrawal, and gradual withdrawal, wherein the dosage of the drug prescribed is reduced or the interval between dosages given is increased. Studies report on the differences in withdrawal strategies of antidiuretic therapy targeted at enuresis in pediatric populations. Several studies have reported on the application of structured withdrawal of desmopressin, indicating that gradual withdrawal of desmopressin therapy results in prolonged intervals of continence without relapse. However, to the best of our knowledge, no studies have investigated the strategy of withdrawal of pharmacological treatment with solifenacin and/or mirabegron in children diagnosed with urinary incontinence that have achieved continence on these pharmaceuticals. Our study is proposed to ensure an evidence-based approach to a withdrawal of strategy for pharmacological treatment with solifenacin and/or mirabegron in children with urinary incontinence.

Objectives: The primary objective is to investigate if abrupt withdrawal versus gradual withdrawal of pharmacotherapy (solifenacin and/or mirabegron) influences the risk of recurrence of incontinence. We hypothesize that gradual withdrawal is superior to abrupt withdrawal regarding the risk of recurrence of incontinence.

Study design: This is an open-label prospective randomized trial, allocating participant to each of the three pharmaceutical groups, according to the medical treatment that the child is receiving (solifenacin, mirabegron or solifenacin in combination with mirabegron). Within each pharmaceutical group, the participant will be randomized 1:1 to the intervention being compared; either abrupt withdrawal or gradual withdrawal.

Perspectives:The results are expected to influence the withdrawal strategy of pharmacological treatment with solifenacin and/or mirabegron in children with daytime urinary incontinence.

Ethics: All pharmacological side effects will be handled in accordance with the Danish legislation. No risk or unknown side effects are expected to medical treatment or withdrawal. The therapeutic potential for future patients justifies the project to be carried out. Participation in this study will not lead to any disadvantages for the patient in their treatment. The study will be conducted in accordance with the protocol, applicable regulatory requirements according to Good Clinical Practice and the ethical principles of the Declaration of Helsinki. The study has been approved by the authorities and was initiated in May 2024. Significant additions or changes to the protocol may be conducted after the application for amendment is approved by the Regulatory Authority and the Ethics Committee. Information regarding the participants is protected according to the General Data Protection Regulation and the actual law. The study is registered at the research inventory of the Regions of Denmark (1-16-02-211-24) and at Aarhus University (ARG-2024-731-23833). The study is registered at CTIS (EU CT 2023-510187-13-00).

ELIGIBILITY:
Inclusion Criteria:

1. The participants custody holder(s) must voluntarily sign and date an informed consent prior to initiation of any study specific procedures.
2. Age 5 to 14 years (inclusive) at the time of signing the consent and inclusion.
3. Diagnose with urinary incontinence as per ICCS criteria.
4. Pharmacological treatment with solifenacin and/or mirabegron.
5. Continence has been achieved on pharmacological therapy with solifenacin and/or mirabegron.
6. Previously withdrawal attempts are accepted.
7. Continence remained on the same dosage of medication for a minimum of three months.

Exclusion Criteria:

1. Inability of the patent(s) or parental custody holder(s) to understand the Danish written and oral information.
2. Neurogenic detrusor overactivity (neurogenic bladder)

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 216 (Estimated)
Dates: Start 2024-05-27 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Recurrence of incontinence after withdrawal | Baseline and up to 12 months follow-up
  Assessed by a 14-day calendar of incontinence episodes

SECONDARY OUTCOMES:
Development of any symptoms related to abrupt or gradual withdrawal symptoms | Baseline up to 44 days after initiation of withdrawal
  Assessed by a questionnaire on withdrawal symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Luise Borch, MD, PhD, Study Director — Department of Pediatric and Adolescent Medicine, Gødstrup Hospital
Locations (5):
- Denmark (5):
  - Department of Pediatric and Adolescent Medicine, Aalborg University Hospital, Aalborg, Aalborg
  - Department of Pediatric and Adolescent Medicine, Aarhus University Hospital, Aarhus, Aarhus N
  - Department of Pediatric and Adolescent medicine, Esbjerg Hospital, Esbjerg, Esbjerg
  - Department of Pediatric and Adolescent Medicine, Gødstrup Hospital, Herning, Herning
  - Department of Pediatric and Adolescent Medicine, Kolding Hospital, Kolding, Kolding

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Svendsen AM, Hagstrom S, Kamperis K, Andersen AE, Henneberg NC, Van Batavia J, Olesen AE, Borch L. Strategy for Withdrawal of Pharmacological Treatment for Urinary Incontinence in Children (StayDry): Protocol for an Open-Label Prospective Randomized Trial. JMIR Res Protoc. 2025 Jul 9;14:e63226. doi: 10.2196/63226. PMID 40633093